CLINICAL TRIAL: NCT06743529
Title: Immediate Versus Substantiated Antibiotic Therapy in Suspected Non-Severe Ventilator-Associated Pneumonia: A Randomized Controlled Trial
Brief Title: Immediate Versus Substantiated Antibiotic Therapy in Suspected Non-Severe Ventilator-Associated Pneumonia
Acronym: POSTPONE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC24_0466
Record Dates: First submitted 2024-12-10; First posted 2024-12-20 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Ventilator-Associated Pneumonia (VAP)
Keywords: Intensive care medicine; Intensive care; Ventilator-associated pneumonia; antibiotic sparing
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate strategy (Active Comparator): Usual Care
  Interventions: Procedure: control group
- Conservative strategy (Experimental): Conservative strategy
  Interventions: Procedure: Conservative strategy

INTERVENTIONS:
Procedure: control group — immediate empiric Antibiotic Therapy (started within 1 hour after randomization) with antibiotic(s) chosen by the bedside physician based on time of ventilator-associated pneumoniaoccurrence, risk of antimicrobial resistance, local ecology, and local protocol. If the respiratory samples are negative, Antibiotic Therapy will be stopped. If ventilator-associated pneumonia is confirmed by positive samples, Antibiotic Therapy active against the recovered bacterial specie(s) will be given for a total of 7 days.
  Arms: Immediate strategy
Procedure: Conservative strategy — No Antibiotic Therapy until receipt of the respiratory sample culture and/or polymerase chain reaction results. If these results are negative, no Antibiotic Therapy is given. If they are positive (confirmed ventilator-associated pneumonia), Antibiotic Therapy is started as appropriate for the bacterial specie(s) detected by culture and/or polymerase chain reaction, without considering gram-stain results and without waiting for antimicrobial susceptibility testing results, and continued for a total of 7 days of Antibiotic Therapy active against the identified bacterial specie(s).
  Arms: Conservative strategy

SUMMARY:
Ventilator-associated pneumonia is the leading nosocomial infection in the intensive care units, and is associated with prolonged mechanical ventilation and overuse of antibiotics. Initiating antibiotic therapy immediately after bacteriological sampling (immediate strategy) may expose uninfected patients to unnecessary treatment, while waiting for bacteriological confirmation (conservative strategy) may delay ventilator-associated pneumonia in infected patients.

The decision to start antibiotic therapy for ventilator-associated pneumonia takes three points into account: diagnostic probability, the risks to the patient if Antibiotic Therapy is delayed, and the risk of selection of resistant bacteria. Diagnostic probability is limited, given the subjective and non-specific nature of the diagnostic criteria, and only 30-50% of suspected cases are confirmed bacteriologically (whereas samples are only taken when the pre-test probability is sufficient). The risks associated with delayed antibiotic therapy are unknown, as few observational studies have directly assessed the impact of the timing of Antibiotic Therapy initiation on outcome (frequent confusion between delayed and inappropriate Antibiotic Therapy).

Iregui et al. found that delaying Antibiotic Therapy by more than 24 hours was associated with higher mortality. However, more recent before-and-after studies have shown that the conservative strategy was associated with lower mortality, more frequently appropriate initial Antibiotic Therapy and shorter duration of Antibiotic Therapy. Similarly, in a recent before-and-after study by our team, initiating antibiotic therapy only upon microbiological confirmation of ventilator-associated pneumonia without septic shock or severe acute respiratory distress syndrome was not associated with an increase in ventilation time, length of stay or excess mortality at D28; but was associated with antibiotic therapy that was more often appropriate (DELAVAP, MARTIN et al, Annals of Intensive Care, 2024). Finally, the recent multicenter TARPP pilot study in surgical intensive care suggests that antibiotic therapy initiated on the basis of microbiological data in patients with suspected ventilator-associated pneumonia not requiring vasopressor support is not associated with a poorer outcome than immediate antibiotic therapy without documentation (the only randomized study on this subject).

Antibiotic Therapy for suspected ventilator-associated pneumonia that is not subsequently confirmed is an unnecessary use of antibiotics and carries a risk of selection of resistant bacteria, with adverse effects on public health. It has been reported that a conservative Antibiotic Therapy prescription strategy for intensive care units -acquired infections reduces Antibiotic Therapy use and the incidence of acquired β-lactamase-producing Enterobacteriaceae infections.

Overall, in patients with suspected ventilator-associated pneumonia but no signs of clinical severity, given the uncertainty about attributable mortality and concerns about bacterial resistance, the evaluation of the conservative Antibiotic Therapy strategy is reasonable. Some French intensive care units already delay Antibiotic Therapy until confirmation of ventilator-associated pneumonia, except in patients with severe hypoxemia or the need for vasopressor support.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation for longer than 48 hours
* Respiratory sample collection taken less than two hours ago (at physician discretion, according to local protocol) for a first episode of suspected ventilator-associated pneumonia (meeting the following prespecified criteria) :

  * new or changing chest X-ray infiltrates
  * plus at least two of the following:

    * body temperature ≥38.5°C or ≤35.5°C,
    * blood leukocyte count >12 000/µL or <4000/µL,
    * purulent tracheobronchial aspirate.
* Age ≥18 years
* Informed consent from the patient or next of kin to participation in the trial, or emergency procedure if no next of kin is available
* Patients affiliated to a social security system

Non-inclusion Criteria:

* Criteria for severe ventilator-associated pneumonia defined as:

  * Vasopressor therapy for onset of septic shock around the time of ventilator-associated pneumonia suspicion
  * Onset or severe worsening of hypoxemia (PaO2/FiO2<150 with 60% FiO2 and 10 mm H2O peak expiratory pressure, or patient on veno-venous extracorporeal membrane oxygenation)
* Immunosuppression defined as :

  * leukocytes <1G/L or neutrophils <0,5 G/L
  * within the last 3 months
  * hematopoietic stem-cell transplant or organ transplant with chronic immunosuppressant therapy
  * HIV infection with CD4<50/mm3
  * chronic corticosteroid use (>0.5 mg/kg day for at least one month within the last three months).
* Patient already on Antibiotic Therapy of predicted duration ≥4 weeks (endocarditis, spondylodiscitis, abscess...)
* Previous ventilator-associated pneumonia suspicion with sampling and/or Antibiotic Therapy for suspected ventilator-associated pneumonia
* Previous inclusion in the trial
* Patient included in an interventional study on ventilator-associated pneumonia management with the same primary endpoint.
* Pregnancy, recent delivery, or breastfeeding
* Correctional facility inmate, adult under guardianship
* Patient under legal protection
* Life expectancy less than 48 hours and/or decision to withhold and/or withdraw life-sustaining therapies
* Organ donor reanimation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2028-12-11 (Estimated); Study Completion 2029-02-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who die whithin 28 days or are still on invasive mechanical ventilation on day 28 | From day 0 to day 28
  To assess, in intensive care units patients with suspected nonsevere ventilator-associated pneumonia (no septic shock or severe acute respiratory distress syndrome), whether delaying antibiotic therapy until ventilator-associated pneumonia is confirmed by a positive respiratory-sample culture and/or polymerase chain reaction test (conservative strategy) neither increases day-28 mortality nor prolongs invasive mechanical ventilation , compared to antibiotic therapy initiation immediately after sampling (immediate strategy).

SECONDARY OUTCOMES:
Sequential Organ Failure Assessment (SOFA) score | From day 0 to day 7
  Daily Sequential Organ Failure Assessment (SOFA)
Modified clinical pulmonary infection score (mCPIS) | From day 0 to day 7
  Daily mcPIS
Clinical cure | day 7
  Clinical cure is defined as the combination of resolution of signs and symptoms present at enrollment, and improvement or lack of progression of radiological signs
Invasive mechanical ventilation duration | From day 0 to day 28
  Days of invasive mechanical ventilation
Ventilator free days | From day 0 to day 28
Use of vasopressors | From day 0 to day 28
  Days on vasopressors
Use of renal replacement therapy | From day 0 to day 28
  Days on renal replacement therapy
Mortality rates | ICU discharge, an average of 10 days
  ICU discharge mortality rates
Mortality rates | day 28
  Mortality rates at day 28
Mortality rates | day 90
  Mortality rates at day 90
Mortality rates | Hospital discharge, an average of 20 days
  Mortality rates at hospital discharge
ICU stay lenghts | From day 0 until the day of discharge from ICU, an average of 10 days
  ICU stay lenghts (days)
Hospital stay lenghts | From day 0 until the day of discharge from Hospital, an average of 20 days
  Hospital stay lenghts (days)
Incidence of ventilator associated pneumonia related abscess | From day 0 until the day of discharge from ICU, an average of 10 days
Incidence of ventilator associated pneumonia related bacteria | From day 0 until the day of discharge from ICU, an average of 10 days
Incidence and timing of subsequent ventilator associated pneumonia during the hospital stay | From day 0 until the day of discharge from Hospital, an average of 20 days
  Incidence and timing of subsequent ventilator associated pneumonia during the hospital stay: relapse, recurrence, superinfection, ventilator associated pneumonia occurrence after a suspected but refuted ventilator associated pneumonia episode; recurrence is defined as improvements in manifestations (fever, secretions, vasopressor needs, inflammatory biomarkers, and chest radiograph infiltrates) after 7 days' treatment with at least ne antibiotic active on all documented bacteria, followed by the return or worsening of these manifestations with a new respiratory sample (culture, with or without PCR) positive for at least one bacterial species in significant concentrations; the same scenario with a respiratory sample positive for at least one of the initial causative bacteria defined relapse; no improvement in manifestations after 7 days' active treatment with a respiratory sample positive for at least one of the initial causative bacteria defined superinfection.
Incidence of noscomial infections between randomisation and hospital discharge | From day 0 until the day of discharge from Hospital, an average of 20 days
  Nosocomial infections including ventilator asssociated pneumonia, nosocomial pneumonia, bacteremia, catheter-related bloodstream infection, urinary-tract infection, soft-tissue infection, C. difficile infection, and other infections
Incidence of in-hospital nosocomial infections by multiresistant bacteria (MRB) | From day 0 until the day of discharge from Hospital, an average of 20 days
  Defined as any of the following: methicillin-resistant Staphylococcus aureus (MRSA), glycopeptide-intermediate S. aureus (GISA), vancomycin-resistant Enterococcus (VRE), extended-spectrum beta-lactamase-producing Enterobacterales (ESBL-e), carbapenemase-producing Enterobacterales (CPE), and imipenem-resistant Acinetobacter baumannii (IRAB).
Incidences of allergies and of diarrhea | From day 0 until the day of discharge from Hospital, an average of 20 days
Antibiotic-free days | day 10
Number of antibotic therapy days by day 28 | day 28
  computed as days of therapy (DOT), defined as the number of days on AT, with each day multiplied by the number of individual antimicrobial agents given on that day, irrespective of the number of doses given.
Broad-spectrum days of therapy (DOT) by day 28 | day 28
  (ceftazidime, piperacillin/tazobactam, cefepime, fluoroquinolones, carbapenems, or new AT for multidrug-resistant Gram-negative bacilli) (number of days on broad-spectrum AT multiplied by the number of individual antimicrobial agents given on each of those days, irrespective of the number of doses given)
Carbapenom days of therapy (DOT) by day 28 | day 28
  Carbapenem DOT by day 28 (number of calendar days during which the patient received at least one carbapenem dose multiplied by the number of individual antimicrobial agents given on each of those days, until day 28, irrespective of the number of doses given).
Ventilator associated pneumonia antibiotic therapy | From day 0 to day 28
  Descriptive data : dual therapy, median time from respiratory sampling to AT, duration, de-escalation (defined as empirical AT stopped or number of empirical antimicrobials decreased or spectrum of empirical AT narrowed, based on AST results)
Descriptive antibiotic therapy data | From day 0 to day 28
  Ventilator associated pneumonia antibiotic therapy: antimicrobial(s), dual therapy, median time from respiratory sampling to antibiotic therapy, duration, de-escalation (defined as empirical AT stopped or number of empirical antimicrobials decreased or spectrum of empirical antibiotic therapy narrowed, based on AST results) , antibiotic therapy for reasons other than suspected VAP: antimicrobial, duration, reason
Descriptive bacteriological data | From day 0 to day 28
  gram stain, organisms recovered (cultured and/or identified by PCR), and antimicrobial resistance profiles
Descriptive clinical, laboratory and radiological data 48 hours before ventilator associated pneumonia suspicion | 48 hours before ventilator asociated pneumonia suspicion
Proportion of patients with confirmed ventilator associated pneumonia | From day 0 to day 28
Number of patients given active/inactive/unnecessary antibiotic therapy on day 0 and on the day of antibiotic therapy initiation | Day 0 and on the day of antibiotic therapy initiation, an average of 1 day
  Number of patients given active/inactive/unnecessary antibiotic therapy on day 0 and on the day of antibiotic therapy initiation (with active defined as at least one antimicrobial agent active against each bacterial species isolated from respiratory samples in concentrations greater than prespecified thresholds, based on AST; inactive defined as not meeting criteria for active AT; and unnecessary defined as antibiotic therapy given before sample results with these being negative)
Number of patients with suitable antibotic therapy (defined as active antibiotic therapy or spared antibiotic therapy as defined below) on day 0 and on the day of antibiotic therapy initiation in the conservative strategy arm | Day 0 and on the day of antibiotic therapy initiation, until discharge from intensive care unit or up to 28 days
  * Number of patients given substantiated antibotic therapy defined as started upon receipt of positive respiratory-sample culture and/or PCR test results
  * Number of patients given rescue antibotic therapy defined as started, in a conservative group patient, after sampling but before culture and/or PCR results, due to the development of ventilator associated pneumonia severity criteria (shock or severe ARDS)
  * Number of patients spared antibotic therapy for the suspected ventilator associated pneumonia episode, that is, not given antibotic therapy after sampling and having negative respiratory-sample results
Incremental cost-utility ratio (ICUR) | day 90
  The incremental cost-utility ratio (ICUR, cost per quality-adjusted life year [QALY] gained) of the two strategies will be computed from a collective perspective and with a 90-day time horizon then compared between the two groups.

OTHER OUTCOMES:
Cost-utility analysis (CUA) | day 90
  To determine whether, in patients who have suspected non-severe VAP (no septic shock or severe ARDS), postponing AT until VAP is confirmed (by a positive respiratory-sample culture and/or PCR) is cost-efficient, compared to the immediate strategy, from a collective perspective (considering costs to the National Health Insurance (NHI) system and hospital) and with a 90-day time horizon. A cost-utility analysis (CUA) will be performed.
  The effectiveness of the two compared strategies will be assessed in terms of potential changes in quality of life and survival (CUA).c.
EQ-5D-5L EuroQol score | day 0
  Quality of life will be assessed using the EQ5D EuroQol score
EQ-5D-5L EuroQol score | day 28
  Quality of life will be assessed using the EQ5D-5L EuroQol score
EQ-5D-5L EuroQol score | day 90
  Quality of life will be assessed using the EQ5D-5L EuroQol score

CONTACTS AND LOCATIONS:
Locations (40):
- France (39):
  - CHU Angers, Angers, France
  - CH Angoulème, Angoulème, France
  - CH Argenteuil, Argenteuil, France
  - CHU Nantes, Nantes, France
  - CH d'Arles, Arles
  - CH Avignon, Avignon
  - Hôpital Nord Franche Comté, Belfort
  - CHU de Bordeaux, Bordeaux
  - CH Simone Veil, Cannes
  - CH Public du Cotentin, Cherbourg
  - CH Cholet, Cholet
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CH Dax, Dax
  - CHU Dijon, Dijon
  - APHP - Hôpital Raymond Poincaré, Garches
  - CHD Vendée, La Roche-sur-Yon
  - CH Versailles, Le Chesnay
  - CH Le Mans, Le Mans
  - CH Emile Roux, Le Puy-en-Velay
  - CHRU Lille, Lille
  - GHB Sud- Hôpital de Lorient, Lorient
  - CHU de Lyon - Hôpital Edouard Herriot, Lyon
  - CH de Melun, Melun
  - CH de Mont de Marsan, Mont-de-Marsan
  - CHU Nice -Hôpital Pasteur, Nice
  - CHU Nice - Hôpital de l'Archet, Nice
  - CHR d'Orléans, Orléans
  - APHP - Hôpital Cochin, Paris
  - APHP - Hôpital Tenon, Paris
  - CH de Pau, Pau
  - CHU Rennes, Rennes
  - CH de Saint-Nazaire, Saint-Nazaire
  - CH de Saint-Malo, St-Malo
  - CHRU de Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - CHRU de Strasbourg -Hôpital de Hautepierre, Strasbourg
  - Hôpital Foch, Suresnes
  - CHRU De Tours, Tours
  - CH de Valenciennes, Valenciennes
  - CH Bretagne Atlantique, Vannes
- CHU La Guadeloupe, Pointe-à-Pitre, Guadeloupe